CLINICAL TRIAL: NCT03950388
Title: A Cluster Randomised Controlled Trial of a Ward-Based Intervention to Improve Access to Psychologically-Informed Care and Psychological Therapy for Mental Health In-Patients
Brief Title: Trial of a Ward-Based Intervention to Improve Access to Psychologically-Informed Care and Psychological Therapy for Mental Health In-Patients
Acronym: TULIPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manchester (Other)
Collaborators: Clinical Trials Unit, Manchester (Other)
Responsible Party: Principal Investigator, Dr Katherine Berry, Senior Lecturer in Clinical Psychology, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R122297
Record Dates: First submitted 2019-04-18; First posted 2019-05-15 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (No Intervention)
- Intervention (Experimental)
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Wards randomly assigned to receive the intervention will have a Band 8a Psychologist based on the ward for 0.5FTE for 7 months. During this time, all patients will be involved with the proposed stepped model of care intervention at one of three levels. The level the patient receives will be decided by the multidisciplinary ward team. At Step one, all patients will have a psychological formulation developed by the psychologist in conjunction with the patient or members of the ward team. At Step 2, all qualified nurses will be trained and supervised to deliver guided self-help material of psychological interventions targeting key problem areas for patients. At Step 3, patients will be offered up to 16, one-to-one therapy sessions with the psychologist.
  Arms: Intervention

SUMMARY:
The Care Quality Commission (2017) concludes that too often care for people with severe mental health problems on mental health inpatient wards institutionalises people, rather than helping them to have an independent life in the community. There is good evidence that psychological interventions improve patient well-being and independent living, but patients on acute mental health wards often do not have access to evidence-based psychological therapies which are strongly advised by NICE guidance for severe mental health problems (e.g. NICE, 2011). The overall aim of this programme of work is to increase patient access to psychological therapies on acute mental health inpatient wards. Stage one of the programme aimed to identify barriers and facilitators to delivering therapy in these settings through a large qualitative study. The key output of stage one was an intervention protocol that is designed to be delivered on acute wards to increase patient access to psychologically-informed care and therapy. Stage two of the programme aims to test the effects of the intervention on patient wellbeing and serious incidents on the ward which are routinely collated by wards and patient and staff contact is not required (primary outcomes), patient social functioning and symptoms, staff burnout, ward atmosphere from staff and patient perspectives and cost effectiveness of the intervention (secondary outcomes). The study is a single blind, pragmatic, cluster randomised controlled trial and will recruit thirty-four wards across England that will be randomised to receive the new intervention plus treatment as usual, or treatment as usual only. Primary and secondary outcomes will be assessed at baseline and 6-month and 9-month follow-ups, with serious incidents on the ward collected at an additional 3-month follow-up. A process evaluation will be nested within the trial to understand factors that influence the effects of the intervention and implementation in real world settings.

ELIGIBILITY:
Inclusion Criteria:

Ward:

1) Generic, working-age, adult acute mental health wards.

Staff (RCT Outcome Measures):

1. Consent to complete self-report measures.
2. Based on the ward for at least 75% of their working week.

Patient (RCT Outcome Measures):

1. Capacity to consent to complete the self-report measures
2. Sufficient levels of concentration to complete the required battery of self-report measures with breaks if needed. This will be determined by the researcher when meeting the participant and in collaboration with the clinical team.
3. Sufficient English language proficiency to take part in qualitative interviews or agreement to the use of an interpreter. This will be determined by the researcher when meeting the participant and in collaboration with the clinical team.

Staff (Semi-structured interviews):

1. Consent to have interviews digitally audio recorded.
2. Direct experience of working with patients with severe mental health problems on an acute inpatient ward that has taken part in the RCT.

Patients (Semi-structured interviews):

1. Capacity to provide informed consent for interviews.
2. Consent to have interviews recorded.
3. At least one week's experience of being an in-patient on an acute in-patient ward that has taken part in the RCT.
4. Sufficient English language proficiency to take part in qualitative interviews or agreement to the use of an interpreter.

Exclusion Criteria:

Ward:

1. Wards that have a specialist function, such as older people, intensive care or rehabilitation.
2. Wards that already have more than 1 session of dedicated psychological therapy input per week. This is because we need to ensure treatment as usual does not include significant elements of the intervention we are aiming to test.

Staff (RCT Outcome Measures):

1. Non-permanent staff, such as bank or agency workers.
2. Staff who are planning to leave the ward before the intervention period starts.

Patient (RCT Outcome Measures):

1. Patients whose discharge is planned for before the start of the intervention period.
2. Unable to complete self-report measures due to difficulties with concentration or high levels of distress. This will be determined by the researcher when meeting the participant and in collaboration with the clinical team.
3. Unable or unwilling to provide informed consent.

Staff (Semi-structured interviews):

1. Non-permanent staff, such as bank or agency workers.
2. Working on the ward for less than 2 weeks at the time of the interview.
3. Unwilling to consent to having interviews audio recorded.

Patient (Semi-structured interviews):

1. Less than one week's experience of in-patient care at the time of the interview.
2. Unable or unwilling to provide informed consent for interviews.
3. Unable or unwilling to have interviews audio recorded.
4. Insufficient English language proficiency to take part in the interview and does not consent to the use of an interpreter.
5. Insufficient English language proficiency to complete the self-report measures and does not consent to the use of an interpreter.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2019-10-21 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Patient wellbeing | Baseline, 6 months and 9 months
  Patient well being using the Warwick-Edinburgh Mental Well-being Questionnaire. WEMWBS: Scale: 1= None of the time, 2 = Rarely, 3 = Some of the time, 4 = Often, 5 = All of the time. Participants are asked to select an option considering the statement over the past 2 weeks. WEMWBS is a 14 item scale with 5 response categories, summed to provide a single score ranging from 14-70. The items are all worded positively and cover both feeling and functioning aspects of mental wellbeing, thereby making the concept more accessible.
Serious incidents on ward | Baseline, 3 months, 6 months and 9 months
  Report taken from each Trust about the number of different serious incidents reported on a ward across a 3 month time period. Serious Incidents: Taken from current reports pulled by each trust to monitor the number of incidents which occur within a ward. Categorised by each Trust using a levelling system of 1-5 with 5 being the most serious level. The incidents are also categorised by event type which varies at each Trust and again is the responsibility of each data entry personnel to assign a category. Data to be taken at baseline for the 3 months prior, at 3 months for the 3 months prior, at 6 months for the 3 months prior and at 9 months for the 3 months prior

SECONDARY OUTCOMES:
Whether the intervention improves patients' symptoms | Baseline, 6 months and 9 months
  Using Brief Symptom Inventory questionnaire. Scale: 0= Not at all; 1 = a little bit, 2 = moderately, 3= quite a bit, 4 = extremely, R= refused Duration: answers based on past 7 days including day of completion Score: The items are all worded positively and cover both feeling and functioning aspects of mental wellbeing.Respondents rank each feeling item (e.g., "your feelings being easily hurt") on a 5-point scale ranging from 0 (not at all) to 4 (extremely). Rankings characterize the intensity of distress during the past seven days.
  The items comprising each of the 9 primary symptom dimensions are as follows:
  * Somatization: Items 2, 7, 23, 29, 30, 33, and 37
  * Obsession-Compulsion: Items 5, 15, 26, 27, 32, and 36
  * Interpersonal Sensitivity: Items 20, 21, 22, and 42
  * Depression: Items 9, 16, 17, 18, 35, and 50
  * Anxiety: Items 1, 12, 19, 38, 45, and 49
  * Hostility: Items 6, 13, 40, 41, and 46
  * Phobic Anxiety: Items 8, 28, 31, 43, and 47
  * Paranoid Ideation: Items
Whether the intervention improves staff perceptions of ward atmosphere. | 6 months
  Using the VOTE Scale: Strongly agree, agree, slightly agree, slightly disagree, disagree, strongly disagree
Whether the intervention improves patient perceptions of ward atmosphere. | 6 months
  Using the VOICE Scale: Strongly agree, agree, slightly agree, slightly disagree, disagree, strongly disagree
Whether the intervention reduces staff burnout. | Baseline, 6 months and 9 months
  Using Maslach Burnout Inventory questionnaire
  MBI:
  Scale:0 = Never, 1 = a few times a year or less, 2 = once a more or less, 3= a few times a month, 4 = once a week, 5 = a few times a week, 6 = every day.
  Duration: Based on 22 statements the participant is to note from 0-6 next to the statement that bests describes how frequently they feel that way.
  Score: The participants receive an emotional exhaustion score (EE) (Qs 1,2,3,6,8,13,14,16,20). A depersonalization score (Dep) (Qs 5,10,11,15,22) A professional accomplishment score (PA) (Qs 4,7,9,12,17,18,19,21). EE score is High (27 or over), Moderate (17-26) and low (0-16). Dep score is high (13 or over), Moderate (7-12) or Low (0-6). PA score is high (39 or over), moderate (32-38) or low (0-31).
Cost-effectiveness of the psychological service model using health economic measures. | Baseline, 6 months and 9 months
  Using Health Economics measures (using service use questionnaires) Service use inventory developed from CSRI.
Identify contextual factors that promote/inhibit implementation and routine incorporation of psychologically-informed care and therapies into everyday practice. | 6 months
  Using implementation fidelity data from the psychologist and ward nurses
Identify contextual factors that promote/inhibit implementation and routine incorporation of psychologically-informed care and therapies into everyday practice. | 6 months
  Using observation data - observe 6 chosen intervention wards
Identify contextual factors that promote/inhibit implementation and routine incorporation of psychologically-informed care and therapies into everyday practice. | 6 months
  Using interview data - interviews with patients and staff on intervention wards
Whether the intervention improves social functioning. | Baseline, 6 months and 9 months
  Using Personal and Social Performance Scale. One for the a-c areas and one specific to the d area.
  Degrees of severity areas a-c. Degrees of severity area d. Absent, Mild, Manifest, Marked, Severe, Very Severe. Overall score of between 0-100 to be given based on the scores for each of the areas (a-d)
Improves quality of life | Baseline, 6 months and 9 months
  EQ-5D-5L:
  Each of the 5 dimensions comprising the EQ-5D descriptive system is divided into 5 levels of perceived problems:
  Level 1: indicating no problem Level 2: indicating slight problems Level 3: indicating moderate problems Level 4: indicating severe problems Level 5: indicating extreme problems A unique health state is defined by combining 1 level from each of the 5 dimensions.
  Scoring: level 1 is coded as 1, level 2 as 2, level 3 as 3, level 4 as 4 and level 5 as 5. There should be only ONE response for each dimension NB: Missing values can be coded as '9'.NB: Ambiguous values (e.g. 2 boxes are ticked for a single dimension) should be treated as missing values. The EQ VAS should be coded as per where the X is placed on a scale of 0-100 with 100= the best health and 0= the worst health. Missing values should be coded as '999'.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Greater Manchester Mental Health NHS Foundation Trust, Manchester, Greater Manchester
  - Leed & York Partnership NHS Foundation Trust, Leeds

REFERENCES:
- [Derived] Johnston I, Edge D, Wilson P, Beinaraviciute A, Bucci S, Drake R, Gilworth G, Haddock G, Handerer F, Kaur S, Lovell K, Morley H, Price O, Samji M, Berry K. Increasing access to psychological therapy on acute mental health wards: staff and patient experiences of a stepped psychological intervention. BMC Psychiatry. 2025 Mar 28;25(1):300. doi: 10.1186/s12888-025-06721-7. PMID 40155872
- [Derived] Berry K, Raphael J, Wilson H, Bucci S, Drake RJ, Edge D, Emsley R, Gilworth G, Lovell K, Odebiyi B, Price O, Sutton M, Winter R, Haddock G. A cluster randomised controlled trial of a ward-based intervention to improve access to psychologically-informed care and psychological therapy for mental health in-patients. BMC Psychiatry. 2022 Feb 3;22(1):82. doi: 10.1186/s12888-022-03696-7. PMID 35114980